CLINICAL TRIAL: NCT06909500
Title: ACT on Vaping: Digital Therapeutic for Young Adult Vaping Cessation
Brief Title: A Digital Intervention (ACT on Vaping App) for Vaping Cessation in Young Adult E-Cigarette Users
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1125194; NCI-2025-01611 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UH3DA057032 (NIH)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-04

CONDITIONS: Nicotine Dependence; Tobacco-Related Carcinoma
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The control app will also be called ACT on Vaping in participant-facing materials, for blinding purposes; Any outcome evaluator who has direct contact with participants will remain blinded to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (ACT on Vaping app (Version A) + incentivized texts + intervention texts) (Experimental): Participants receive access to the ACT on Vaping app utilizing Acceptance and Commitment Therapy. Participants also receive text message intervention content, as well as incentivized text message check-ins at 2 weeks, 2 months, and 4 months to assess changes in vaping on study.
  Interventions: Behavioral: Smartphone app; Other: Text Message; Other: Survey Administration
- Arm II (ACT on Vaping app (Version B) + incentivized texts) (Sham Comparator): Participants receive access to the ACT on Vaping app including health education content. Participants receive incentivized text message check-ins at 2 weeks, 2 months, and 4 months to assess changes in vaping on study.
  Interventions: Behavioral: Smartphone app; Other: Text Message; Other: Survey Administration

INTERVENTIONS:
Behavioral: Smartphone app — Receive access to the ACT on Vaping app
  Other Names: ACT on Vaping (Version A)
  Arms: Arm I (ACT on Vaping app (Version A) + incentivized texts + intervention texts)
Behavioral: Smartphone app — Receive access to the ACT on Vaping app
  Other Names: ACT on Vaping (Version B)
  Arms: Arm II (ACT on Vaping app (Version B) + incentivized texts)
Other: Text Message — Receive incentivized text messages to access vaping status
  Other Names: SMS Text
Other: Text Message — Receive intervention text messages
  Other Names: SMS Text
  Arms: Arm I (ACT on Vaping app (Version A) + incentivized texts + intervention texts)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a smartphone application (app) called Acceptance and Commitment Therapy (ACT) on Vaping for helping young adults quit using electronic cigarettes (e-cigarettes). E-cigarettes pose numerous risks, particularly to youth and young adults. Addressing the high prevalence of e-cigarette use by young adults requires effective and accessible treatments to support current users to quit. Research shows this group prefers and benefits from newer methods of treatment delivery such as digital interventions. ACT on Vaping is a digital therapeutic intended to deliver behavioral therapy to young adults who vape to motivate and support abstinence from all nicotine and tobacco products. The app contains sessions that promote awareness of cues that trigger tobacco use and teach skills for responding to these triggers in a way that is tailored for the participant's readiness to quit. Receiving access to the ACT on Vaping app may be effective in helping young adults quit vaping.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants use the ACT on Vaping app (Version A) and receive a text messaging program to motivate and support quitting. Participants also receive incentivized text message check-ins at 2 weeks, 2 months, and 4 months to assess their vaping status.

ARM II: Participants use the ACT on Vaping app (Version B) and receive incentivized text message check-ins at 2 weeks, 2 months, and 4 months to assess their vaping status.

After completion of study intervention, participants are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Age of majority (to provide informed consent) in current state/territory of residence
* Current weekly user of e-cigarette product(s) for the last 30 days
* Has a smartphone; either an Android (running version 12 or higher) or iPhone (running iOS version 17 or higher, iPhone 11 or more recent)
* Experience downloading and using one or more apps on their smartphone
* Have a mobile data plan and/or access to WiFi to support the use of the ACT on Vaping app
* Has access to text messaging
* Has an email address
* United States (US) resident, with a US mailing address
* Willing to complete all study procedures
* Comfortable reading and writing in English

Exclusion Criteria:

* Currently using other tobacco cessation treatments at the time of screening, including pharmacotherapy or behavioral support (note: use of these treatment is allowable during trial participation)
* Member of the same household as another research participant
* Currently in prison
* Google voice number as sole phone number, due to its association with fraudulent study entry attempts
* Is ineligible per fraud prevention protocol
* Employees/family of investigator or study center

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1372 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Cotinine-confirmed 7-day point prevalence abstinence from all nicotine and tobacco | At 6 months post-randomization
  Biochemically confirmed 7-day abstinence from all nicotine and tobacco (excluding FDA-approved pharmacotherapies).

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence from all nicotine and tobacco | At 6 months post-randomization
  Proportion of participants self-reporting 7-day abstinence from all nicotine and tobacco (excluding FDA-approved pharmacotherapies).
Self-reported 7-day point prevalence abstinence from all nicotine and tobacco | At 3 months post-randomization
  Proportion of participants self-reporting 7-day abstinence from all nicotine and tobacco (excluding FDA-approved pharmacotherapies).
Cotinine-confirmed 7-day point prevalence abstinence from all nicotine and tobacco | 3 At 3 months post-randomization
  Biochemically-confirmed 7-day abstinence from all nicotine and tobacco (excluding FDA-approved pharmacotherapies).
Self-reported 30-day point prevalence abstinence from all nicotine and tobacco | At 3 months post-randomization
  Proportion of participants self-reporting 30-day abstinence from all nicotine and tobacco (including FDA-approved pharmacotherapies).
Self-reported 30-day point prevalence abstinence from all nicotine and tobacco | At 6 months post-randomization
  Proportion of participants self-reporting 30-day abstinence from all nicotine and tobacco (including FDA-approved pharmacotherapies).
Self-reported 7-day point prevalence abstinence from vaping | At 3 months post-randomization
  Proportion of participants self-reporting 7-day abstinence from vaping.
Self-reported 30-day point prevalence abstinence from vaping | At 3 months post-randomization
  Proportion of participants self-reporting 30-day abstinence from vaping.
Self-reported 7-day point prevalence abstinence from vaping | At 6 months post-randomization
  Proportion of participants self-reporting 7-day abstinence from vaping.
Self-reported 30-day point prevalence abstinence from vaping | At 6 months post-randomization
  Proportion of participants self-reporting 30-day abstinence from vaping.
Number of 24-hour quit attempts | Baseline to 3 months post-randomization
  Number of times between baseline and 3-month follow-up that participant stopped using all nicotine and tobacco (excluding FDA-approved pharmacotherapies) for 24 hours or longer.
Prolonged self-reported abstinence from all nicotine and tobacco for 90 days | At 6 months post-randomization
  Proportion of participants self-reporting no nicotine or tobacco use (excluding FDA-approved pharmacotherapies) for 90 days prior to 6-month follow-up.
Change in readiness to quit using electronic cigarettes (e-cigarettes) on the Contemplation Ladder | Baseline to 3 months post-randomization
  Self-reported motivation to quit smoking e-cigarettes (Contemplation Ladder), rated 1-10. Higher scores indicate greater motivation to quit [i.e., high (>5) vs. low (5 or less)].

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to preserve & share the following scientific data:
  * Survey Data: De-identified individual & aggregate survey data (including raw and recoded data) necessary to replicate main outcomes will be shared
  * App utilization data: Individual level, de-identified aggregate data necessary to replicate main outcomes will be shared
  Documentation made publicly available to the research community will also include PDFs of the following:
  * Survey instruments with proprietary measures redacted
  * A description of the data collection methods
  * Copies of study consent forms & other relevant documentation of IRB approval & limitations on data sharing or usage
  * Survey codebook
  * Methods used to code or summarize open-text survey responses
  * Steps taken to remove direct & indirect identifiers in the data
  * Description of the software & analytical methods used in survey data analyses
  * Code used in data analyses
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Final data submission and release of data used in publications will occur at the time of publication. Other shared data will be made available at or before the end of the project period. We will follow the data retention plan of the final selected repository, but at a minimum, we intend to ensure that data is available for a period of not less than 5 years after the end of this trial.
Access Criteria: All data sharing will be done in compliance with NIH data sharing policies, applicable laws and regulations, and in accordance with guidance from journal publishers. At this time, we plan to share scientific data and meta-data in NCI's Cancer Data Service (CDS). CDS allows open and controlled access to data to ensure access is provided to qualified researchers, data access is tracked, and users understand how to cite and credit use of the data. Data will only be shared for non-profit, non-commercial and non-proprietary purposes to qualified researchers or as allowed by CDS. Based on the nature of the data, which is not sensitive, we anticipate making it publicly available (as opposed to controlled access) but will follow final recommendations from the IRB as to whether access should be controlled.
URL: https://dataservice.datacommons.cancer.gov/#/home